CLINICAL TRIAL: NCT01140399
Title: Impact of Different Therapeutic Approaches in Patients With Cardiorenal Syndrome in the Setting of Acute Decompensated Congestive Heart Failure (ADCHF)
Brief Title: REWORD-HF REverse WOrsening Renal Function in Decompensated Heart Failure
Acronym: REWORD-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Niguarda Hospital (Other)
Collaborators: Associazione Nazionale Medici Cardiologi Ospedalieri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT code 2009-014; FO001
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: 1 Acute Decompensated Heart Failure; 2 Cardiorenal Syndrome; 3 Ultrafiltration; 4 Dopamine
MeSH Terms: interventions — Furosemide; Dopamine; Ultrafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusional drug treatment (Active Comparator): Diuretics or diuretics plus fixed low dose dopamine infusion
  Interventions: Drug: Furosemide or Furosemide and Dopamine
- Ultrafiltration (Experimental): Device: Ultrafiltration appliance Sessions of 8 h UF are conducted on 2 subsequent days in the first 48 hours after randomization; a third session is performed on day 3 in case of persistent congestion
  Interventions: Device: Ultrafiltration

INTERVENTIONS:
Drug: Furosemide or Furosemide and Dopamine — Patients randomized to pharmacological treatment receive
  * either intravenous diuretics at escalating doses up to 20 mg/h
  * or intravenous diuretics up to 20 mg/h and dopamine infusion at a constant rate of 3 mcg/Kg/m.
  Arms: Infusional drug treatment
Device: Ultrafiltration — All loop diuretics will be discontinued. Rate of fluid removal will be based on the extent of fluid overload as assessed by increase in body weight vs the patient's known dry weight
  * less than 3 kg 200 ml/h
  * more than 3 kg and less than 5 kg 300 mlh
  * more than 5 kg 500 mlh
  Criteria for achievement of target UF goals are removal of > 50% and <70% of fluid excess based on the estimated increase in body weight Diuretic infusion is allowed provided that a minimum of 3 hours after the end of the UF session have elapsed, at a maximum cumulative dose of 100 mg furosemide, till start of the next UF session The use of inotropic agents is prohibited
  Arms: Ultrafiltration

SUMMARY:
The purpose of this study is to determine whether in patients with acute decompensated congestive heart failure and the cardiorenal syndrome, i.e. a state in which therapy directed to improve symptoms is limited by further worsening renal function, fluid removal by ultrafiltration is superior to different pharmacological approaches in acutely relieving congestion and preventing further deterioration in renal function and whether it results in longer admission-free survival 90 days after enrolment

DETAILED DESCRIPTION:
Acute decompensated congestive heart failure (ADCHF), the most common single cause of hospitalization over 65 years, results in 4-8% in-hospital mortality and 30-38% incidence of readmissions within 3 months after discharge. While fluid accumulation remains the main factor causing hospitalization, impaired cardiac output in ADHF causes renal arterial underfilling and increased venous pressure, reducing the glomerular filtration rate and causing acute kidney injury.

Aggressive therapy is required to alleviate volume overload during hospital admission and achievement of a dry weight is capital in preventing rehospitalisation. Currently diuretics are considered the standard of care for volume overload in ADHF, yet any patients, especially those with advanced HF become soon resistant to standard doses of loop diuretics, so escalating doses and the association of thiazides are often required to achieve effective diuresis, an approach that will progressively worsen renal function, causing the cardiorenal syndrome.

When diuretic resistance develops and symptoms persists, mechanical fluid removal via ultrafiltration should be considered. Ultrafiltration is an alternative method of sodium and water removal, that filters plasma water directly across a semipermeable membrane in response to a transmembrane pressure gradient, resulting in an ultrafiltrate that is isoosmotic compared with plasma water, In view of the limits of traditional therapies for the treatment of congestion and concomitant progressive renal dysfunction in ADHF patients, there is a compelling need for additional studies to individuate the better method for fluid removal in volume-overloaded patients and guide management decisions to reduce associated morbidity.

The main objectives of the present project are to evaluate whether in patients with acute decompensated congestive heart failure and the cardiorenal syndrome, i.e. a state in which therapy directed to improve CHF symptoms is limited by further worsening renal function, fluid removal by ultrafiltration is superior to different pharmacological approaches in acutely relieving congestion and preventing further deterioration in renal function and whether it results in longer admission-free survival 90 days after enrolment

ELIGIBILITY:
Inclusion criteria

On admission (screening)

* Informed consent
* Age 18-80 years
* NYHA class III - IV
* Signs of pulmonary (pulmonary rales, and interstitial oedema or pleural effusion on chest Xray) and/or systemic congestion (pitting ankle oedema and enlarged liver or ascites and neck vein distension ≥ 7 cm) and weight gain ≥ 2 kg during the previous week
* Glomerular filtration rate ≥ 30 ml/min
* BNP increased >400 pg/ml (diagnostic cut-off for ADCHF), as confirmatory diagnostic test)

  24 hours after admission (randomization)
* Persistent signs of pulmonary (pulmonary rales, interstitial oedema or pleural effusion on chest Xray) and/or systemic congestion (ankle oedema, enlarged liver or ascites, neck vein distension ≥ 7 cm)
* Serum creatinine or urine output criteria indicative of modified RIFLE (AKI: risk) class at least 1 (increase x 1.5 in serum creatinine or decrease > 25% in GFR or urine output < 0.5 ml/Kg/h for more than 6 hours) 29-30 during diuretic infusion

Exclusion criteria

* Chronic kidney disease stage 4-5 (GFR < 30 ml/min)
* Acute coronary syndromes
* Systolic blood pressure <90 mm Hg/need for intravenous inotropes
* Hematocrit > 45%
* Unattainable venous access
* Contraindications to anticoagulation by heparin
* Systemic infection
* Heart transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Changes in a composite clinical-lab score | Baseline and 96 h after randomization,precisely:48 h after end of the last UF session in the intervention arm;24 h after end of 72 h infusional drug treatment in the control arm
  Changes in a score derived by summing up changes in dyspnea, weight loss, glomerular filtration rate (GFR), brain natriuretic peptide (BNP)

SECONDARY OUTCOMES:
Changes in the dyspnea Likert scale | Measured at day 4, at day 10, at day 90 vs baseline
Changes in modified RIFLE (AKIN) stage | Measured at day 4 vs baseline
Length of stay during index admission | Measured at average day 10
Occurrence of major adverse events | Measured at day 90
  All cause mortality, hospital readmission and unscheduled office and emergency department visits for ADCHF
Days spent alive and out of hospital (DAOH) within 90 days | Measured at day 90
  Sum of days spent alive and out of hospital
BNP changes | Measured at day 0, at day 4, at 10 and day 90
  Changes in BNP at specified times VS baseline
Changes in neutrophil gelatinase associated lipocalin (NGAL) | Measured at day -1, at day 0 and day 4
  Changes in NGAL at specified times VS screening
Changes in Cystatin C (CysC) | Measured at day 0, day 4, day 10 and day 90
  Changes in Cystatin C (CysC) at specified times VS baseline
Treatment-related adverse events | Measured at day 4
  Bleeding, thrombosis, clotting, infection
Adverse changes in blood pressure, heart rate and rhythm | Measured at day 4
  Hypotension (< 90 mmHg), tachycardia (> 110 bpm) arrhythmias
Adverse changes in lab parameters | Measured at day 4
  Hyper-Azotemia (>180 mg/dl), hyper-kaliemia (6.5 mEq/l), hemoconcentration (hematocrit >45%)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Oliva, MD, Study Chair — Heart Failure Heart Transplant Program, Cardiovascular Department, Niguarda Hospital, Milan, Italy; Antonio Santoro, MD, Study Chair — Department of Nephrology, Dialysis and Hypertension, Sant'Orsola Malpighi Hospital, Bologna, Italy
Locations (16):
- Italy (16):
  - Fondazione S. Maugeri. IRCCS Istituto di Cassano Murge, Cassano Murge, Bari
  - Ospedale Civile di Legnano Cardiology, Legnano, Milano
  - Istituto Clinico Humanitas - IRCCS Clinical Cardiology Cardiovascular Department, Rozzano, Milano
  - Azienda Ospedaliera S. Gerardo Heart Failure and Cardiomyopathy Clinic, Monza, Monza Brianza
  - Gruppo Policlinico di Monza Clinical Cardiology and Heart Failure Unit - Cardiology Department, Monza, Monza Brianza
  - Ospedali Riuniti di Ancona Cardiology Presidio Lancisi, Ancona
  - Ospedali Riuniti di Bergamo - Cardiovascular Medicine, Bergamo
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi - Cardiology Unit, Bologna
  - Azienda Ospedaliero-Universitaria di Bologna, Policlinico S.Orsola-Malpighi - Nefrology,Dialysis and Hypertension Unit, Bologna
  - Azienda Ospedaliera Sant'Anna - Cardiology, Como
  - Ospedale SS Annunziata Cardiology, Cosenza
  - Azienda Istituti Ospitalieri di Cremona Cardiology, Cremona
  - Centro Cardiologico Monzino, I.R.C.C.S. Cardiology Intensive Care, Milan
  - Azienda Ospedaliera Niguarda - Heart Failure and Heart Transplant Program, Milan
  - Ospedale Guglielmo da Saliceto Cardiology Department, Piacenza
  - AO Verona Ospedale Civile Maggiore Cardiology Unit, Verona

REFERENCES:
- [Derived] Srivastava M, Harrison N, Caetano AFS, Tan AR, Law M. Ultrafiltration for acute heart failure. Cochrane Database Syst Rev. 2022 Jan 21;1(1):CD013593. doi: 10.1002/14651858.CD013593.pub2. PMID 35061249